CLINICAL TRIAL: NCT03948971
Title: Venous Sinus Pressures in Normal Individuals
Brief Title: Prospective Measurement of Normal Venous Sinus Pressures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00057618
Record Dates: First submitted 2019-05-10; First posted 2019-05-14 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Intracranial Venous Pressures
Keywords: cerebral arteriography

STUDY DESIGN:
Intervention Model Description: Adult patients aged 18-60 years determined to be candidates for elective cerebral arteriography will be screened for inclusion in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Venogram Group (Other): Participants in this group have a scheduled clinically indicated a cerebral angiogram procedure and will undergo a Venogram.
  Interventions: Procedure: Venogram

INTERVENTIONS:
Procedure: Venogram — The 5 French (5F) diagnostic catheter will be navigated into the inferior then superior vena cava and then into the internal jugular bulb on the dominant venous side (as determined from the arteriographic images). Next, a 0.027 inch microcatheter will be navigated using fluoroscopic guidance into the superior sagittal sinus and a venogram will then performed by injecting a small dose of contrast. Next, the venous sinus pressure waveforms will be recorded as the catheter is withdrawn into the jugular bulb and then in the superior vena cava to obtain a central venous pressure. Once completed, the catheters will be removed and the sheaths will be removed. Manual pressure will be held at the venous access site for a few minutes. The arterial sheath will be closed based upon standard arteriogram protocol.

SUMMARY:
The purpose of this research is to document normal intracranial venous sinus pressures. Participants who need to have a cerebral angiogram to evaluate a medical problem not related to Idiopathic Intracranial Hypertension (IIH) will be invited to participate. Participation in this research will not require any extra visits. The intervention will take place in the interventional radiology suite when the subject has an angiogram. IIH is a condition that causes increased pressure in the brain in the absence of a tumor or other diseases that may be causing symptoms. Symptoms include headaches and visual disturbances not explained by other things. In IIH there is a narrowing in the sinuses of the brain that causes the increased pressure.

DETAILED DESCRIPTION:
Patients will be prospectively enrolled into the study. All adult patients, aged of 18-60, determined to be candidates for elective cerebral arteriography will be screened for inclusion in this study. Patients consenting to participate and enrolled in the study will first undergo their standard cerebral angiogram procedure, as clinically indicated. Once the procedure is completed, enrolled subjects will then undergo the study intervention.

1. Insertion of an additional catheter in the femoral vein.
2. Navigation of the catheter into the internal jugular bulb and then catheter navigation into the superior sagittal sinus will result in additional fluoroscopic time (requires ~60 seconds of additional fluoroscopy time; carries a minimum risk of vessel perforation or other untoward event [incidence of complication associated with this procedure in the PI patient series is 0%]). There is additionally some ear pain that can happen with this Venogram.
3. 5-10 minutes of additional procedure time. Much of this time period is merely a waiting period while the pressures stabilize and are recorded.
4. An additional venogram injection through the catheter which exposes subjects to an additional 1-2 ml of contrast dye and 3-4 seconds of additional fluoroscopy time and its associated radiation dose.

ELIGIBILITY:
Inclusion Criteria:

* Candidates for elective cerebral arteriography

Exclusion Criteria:

* All patients with active, or a history of, intracranial venous pathology (arteriovenous malformation, arteriovenous fistulae, idiopathic intracranial hypertension, venous sinus thrombosis).
* Patients with severe daily headaches or symptoms of idiopathic intracranial hypertension will also be excluded.
* Body mass index > 35.
* Known diagnosis of heart failure or pulmonary hypertension.
* Pregnant women will be excluded due to the radiation risk associated with Angiogram and Venogram.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-01-13 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Superior Sagittal Sinus Pressure | during venogram, up to 10 minutes
  Superior sagittal sinus pressure will be recorded in mmHg as the catheter is withdrawn into the jugular bulb.
Torcula Sinus Pressure | during venogram, up to 10 minutes
  Torcula sinus pressure will be recorded in mmHg as the catheter is withdrawn into the jugular bulb.
Dominant Transverse Sinus | during venogram, up to 10 minutes
  Dominant transverse sinus will be recorded in mmHg as the catheter is withdrawn into the jugular bulb.
Dominant Transverse-Sigmoid Sinus Junction | during venogram, up to 10 minutes
  dominant transverse-sigmoid sinus junction will be recorded in mmHg as the catheter is withdrawn into the jugular bulb.
Dominant Sigmoid Sinus | during venogram, up to 10 minutes
  Dominant sigmoid sinus will be recorded in mmHg as the catheter is withdrawn into the jugular bulb.
Dominant Internal Jugular Vein | during venogram, up to 10 minutes
  Dominant internal jugular vein will be recorded in mmHg as the catheter is withdrawn into the jugular bulb.
Central Venous Pressures | during venogram, up to 10 minutes
  Central venous pressures will be recorded in mmHg as the catheter is withdrawn into the jugular bulb.

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Fargen, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Univesity Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No